CLINICAL TRIAL: NCT05526287
Title: Effects of Dual-Task Training on Balance, Gait, Dual-Task Performance, Cognitive Function, Fatigue in People With Multiple Sclerosis
Brief Title: Effects of Dual-Task Training in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Ozkeskin, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOzkeskin
Record Dates: First submitted 2022-07-29; First posted 2022-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Balance; Gait; Dual-Task; Cognitive Function; Functional Mobility; Activities of Daily Living
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-Task Group (Experimental): Participants will receive 8 weeks of dual-task training twice a week and home exercise program.Dual-task training will include motor-motor and motor-cognitive dual-task activities.Home exercise program will include core and lower extremity exercises.Home exercises will be performed three times a week.
  Interventions: Other: Dual-Task Training
- Control Group (Active Comparator): Participants will receive 8 weeks of home exercise program.Home exercise program will include core and lower extremity exercises.Home exercises will be performed three times a week.
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Other: Dual-Task Training — Dual-task training sessions include; walking on treadmill for 10-30 minutes and half of this walking period participants will perform cognitive tasks, cognitive tasks will be repeated on tandem stance position and single leg stance position other half of the session consists of motor-motor dual task activities and gait training on firm and soft surfaces.
  Home exercise program includes lower extremity, core stability and balance exercises and will be performed three times a week.
  Arms: Dual-Task Group
Other: Home Exercise Program — Home exercise program includes lower extremity, core stability and balance exercises and will be performed three times a week.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the effects of dual task training on balance, gait, dual-task performance, cognitive function, fatigue and functional mobility in people with Multiple Sclerosis(MS).

DETAILED DESCRIPTION:
Eligible participants will be randomized to dual-task group or control group. Dual-task group will receive 8 weeks of dual-task training twice a week and home exercise program. Control group will receive only home exercise program for 8 weeks. Each participant will be assessed before and after the 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of MS according to the revised McDonald criteria
* Having Expanded Disability Status Scale score between 0-5.5
* No relapse in the last 30 days
* Having a Mini Mental Test score of 24 and above
* Being fluent in Turkish language
* No condition that prevents exercising

Exclusion Criteria:

* Being pregnant
* Presence of a neuro-musculoskeletal disease other than Multiple Sclerosis
* Having received physiotherapy for balance and gait disorders in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale(BBS) | eight weeks
  BBS, evaluates daily activities including static sitting and standing balance, as well as transfers, turning, and picking up objects from the ground, in 14 items.Scoring is given as 0-4. It scores from 4 (normal performance) to 0 (not able to do the movement) according to the person's ability to do what is asked of them safely and independently. The total score is 56 points. 0-20 indicates high risk, 21-40 indicates medium risk, and 41-64 indicates low risk.
Timed Up And Go Test (TUG) | eight weeks
  It is a frequently used test that evaluates functional mobility and dynamic balance. At the beginning of the test, individuals sit in a chair. A distance of 3 m is set in front of the patient. With the start command, the patient gets up from his seat and walks 3 m, turns around and walks back and sits. With the start command, the time until the moment of sitting on the chair is recorded in seconds.Shorter duration indicates better functional mobility.
Tetrax((Sunlight Medical Ltd, Israel),Computerized Static Posturography Device | eight weeks
  Tetrax (Sunlight Medical Ltd, Israel) computerized posturography device consists of a platform system where data is collected, a computer and software system where data is processed and integrated. Participants will stand on the platform system in 8 different condition. Tetrax will be used to measure static balance and fall risk.

SECONDARY OUTCOMES:
MS Walking Scale-12(MSWS-12) | eight weeks
  MSWS-12 is a 12-item scale evaluating the effect of MS on person's walking ability. MSWS-12 is scored between 12-54. Higher scores indicate more negatively affected walking ability.
Fatigue Severity Index(FSI) | eight weeks
  The scale consists of 9 questions and each question is graded over 7 points.FSI is scored between 0-63. Higher scores indicate more fatigue.
Brief International Cognitive Assesment for MS(BICAMS) | eight weeks
  BICAMS includes Symbol Digit Modalities Test (SDMT), California Verbal Learning Test II (CVLT-II) and Brief Visuospatial Memory Test-Revised (BVMT-R). The total score is determined by summing the scores of the 3 tests. Battery will be used to evaluate cognitive function. Higher scores indicate better cognitive function.
10 Meter Walking Test(10MWT) | eight weeks
  This test calculates the unassisted walking speed of individuals at a distance of 10 meters. In this test, the person will be asked to walk at their normal pace in a pre-measured 10 meter area.
Dual-Task Performance | eight weeks
  Dual-Task performance will be measured with TUG-cognitive and 10MWT-motor. In TUG-cognitive,patient will be counting down by three from a number between 100 and 200 while performing Timed-Up and Go test. In 10MWT-motor,patient will be carrying a tray with 3 water filled 200 ml plastic glasses while walking a 10 m distance.Time will be measured. Longer time to complete task indicates lower dual-task performance.
Dual-Task Questionnaire(DTQ) | eight weeks
  The Dual Task Questionnaire assesses the frequency of difficulties experienced by individuals with neurological injury or disease during activities of daily living that involve dual tasks. DTQ is scored between 0-40. Higher scores indicate more frequent dual-task difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Nur YUCEYAR, MD, Study Chair — Ege University
Locations (1):
- Ege University Faculty of Health Sciences, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No